CLINICAL TRIAL: NCT00877227
Title: Does Folinic Acid Supplementation Decrease Homocysteine Concentrations in Newborns
Brief Title: Does B Vitamin Supplementation Decrease Homocysteine Concentrations in Newborns
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Dr H Blom, clinical biochemical geneticist, Metabolic Unit
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0010-0237
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-04

CONDITIONS: Mild Hyperhomocysteinemia
Keywords: CVA; stroke; newborns; homocysteine; folinic acid
MeSH Terms: conditions — Stroke | interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- folinic acid (Experimental): Folinic acid was given for two weeks as 5-formyltetrahydrofolate (10 mg/ml) (Pharmachemie bv). This solution was administered either intravenously (first week) or orally. To lower homocysteine in adults 5 mg/day folic acid is frequently used. Using an average bodyweight of 70 kg for adults we calculated a daily dose of 70 microgram/kg/day for our newborns
  Interventions: Drug: 5-formyltetrahydrofolate (10 mg/ml) (Pharmachemie bv)
- 2 (No Intervention): control subjects admitted at the Neonatal Intensive Care Unit (NICU)

INTERVENTIONS:
Drug: 5-formyltetrahydrofolate (10 mg/ml) (Pharmachemie bv) — Folinic acid was given for two weeks as 5-formyltetrahydrofolate (10 mg/ml) (Pharmachemie bv). This solution was administered either intravenously (first week) or orally. To lower homocysteine in adults 5 mg/day folic acid is frequently used. Using an average bodyweight of 70 kg for adults we calculated a daily dose of 70 microgram/kg/day for our newborns.
  Other Names: folinic acid
  Arms: folinic acid

SUMMARY:
The purpose of this study is to determine whether supplementation with folinic acid, a B vitamin, lowers the concentrations of total homocysteine in newborns. Increased homocysteine concentrations are associated with an increased risk of cerebrovascular accidents in adult, children and newborns. These increased concentrations can easily and safely be lowered by folic acid in adults.

DETAILED DESCRIPTION:
The incidence of cerebrovascular accidents (CVA) occurring perinatally is relatively high and aspects of the multifactorial pathophysiology remain unclear. Elevated homocysteine concentrations are shown to be associated with an increased risk for CVA in newborns. We want to study the possible homocysteine lowering effect of folinic acid in newborns.

We will include newborns in our prospective randomized folinic acid intervention study from patients admitted to our Neonatal Intensive Care Unit. We will measure total homocysteine (tHcy) and folate concentrations at three time points. The intervention group will be treated with folinic acid (70 µg/kg/day) for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* admitted at our NICU

Exclusion Criteria:

* midline defects
* Extracorporeal membrane oxygenation (ECMO) treatment
* blood transfusion
* overt renal failure

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2003-01; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
lowering total homocysteine concentrations | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henk Blom, Dr, Study Chair — Amsterdam UMC, location VUmc; Marije Hogeveen, MD, Principal Investigator — Radboud University Medical Center Nijmegen
Locations (1):
- Radboud University Medical center Nijmegen, Nijmegen, Netherlands